CLINICAL TRIAL: NCT04582006
Title: Changes of Oral and Intestinal Microbiota After Laparoscopic Sleeve Gastrectomy and Laparoscopic Roux-en-Y Gastric Bypass
Brief Title: Changes of Oral and Intestinal Microbiota After Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Tomasz Stefura, Reasearch Associate, PhD student at 2nd Department of General Surgery, Principal Investigator, Medical Doctor, Jagiellonian University
Other Study IDs: 1072.6120.196.2018-2
Record Dates: First submitted 2020-10-05; First posted 2020-10-09 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LSG: Patients undergoing laparoscopic sleeve gastrectomy.
  Interventions: Procedure: Bariatric surgery
- LRYGB: Patients undergoing laparoscopic Roux-en-Y gastric bypass.
  Interventions: Procedure: Bariatric surgery

INTERVENTIONS:
Procedure: Bariatric surgery — Surgical treatment of morbid obesity.

SUMMARY:
Purpose

The aim of this study was to analyze the changes of microbiota among patients undergoing LSG or LRYGB on two levels of gastrointestinal tract (using oral swab and stool sample). We compared samples from patients before and after bariatric operation.

Materials and methods This prospective cohort study was conducted in one academic, teaching hospital. The recommendations of the Metabolic and Bariatric Surgery Section of the Polish Surgical Society were used as indication for surgery, that is: Body Mass Index (BMI) ≥35 kg/m2 with obesity-related comorbidities or BMI ≥40 kg/m2.

Analysis and endpoints

Primary endpoint was to determine the difference in microbiota present in oral cavity and large intestine between patients before and after bariatric surgery. Secondary endpoint was to compare the difference in microbiota changes between patients undergoing LSG and LRYGB

ELIGIBILITY:
Inclusion Criteria:

* informed consent to participate in the study
* meeting the eligibility criteria for bariatric treatment (either for LSG or LRYGB).

Exclusion Criteria:

* treatment with antibiotics within 30 days prior to gathering microbiological material
* gastrointestinal infections
* inflammatory bowel disease
* thyroid diseases
* cancer (especially the digestive tract)
* immunodeficiency.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The investigators included patients undergoing surgical treatment for morbid obesity.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Change of microbiota in oral cavity | 6 months
Change of microbiota in large intestine | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Department of General Surgery, Jagiellonian University Medical College, Krakow, Małopolska, Poland

IPD SHARING:
Plan to Share IPD: No
We are not planing to share data.

REFERENCES:
- [Derived] Stefura T, Zapala B, Gosiewski T, Skomarovska O, Pedziwiatr M, Major P. Changes in the Composition of Oral and Intestinal Microbiota After Sleeve Gastrectomy and Roux-En-Y Gastric Bypass and Their Impact on Outcomes of Bariatric Surgery. Obes Surg. 2022 May;32(5):1439-1450. doi: 10.1007/s11695-022-05954-9. Epub 2022 Feb 21. PMID 35188608